CLINICAL TRIAL: NCT03514147
Title: The Effect of Pelvic Floor Muscle Training on the Quality of Life and Functionality in Women With Urinary Incontinence: a Randomized Controlled Trial
Brief Title: Pelvic Floor Muscle Training on the Quality of Life in Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0271
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence; Quality of Life
Keywords: Women; Pelvic Floor Muscles
MeSH Terms: conditions — Urinary Incontinence | interventions — Population Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Pelvic Floor Muscle Training in group. Exercise Protocol: The exercise group was supervised and met for 1 hour, one time per week, for 12 weeks. Participants were instructed to perform their respective daily exercises.
  Interventions: Other: Experimental
- Control (Active Comparator): Pelvic Floor Muscle Training in home Exercise Protocol:The same exercise were performed at home for 12 weeks, without supervision. Participants were instructed to perform their respective daily exercises.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — 1. Profile of participants: an anamnesis file was used to collect personal data;
  2. To evaluate the quality of life: To evaluate the quality of life, using International Consultation on Incontinence Questionnaire (ICIQ-Short form) in women with urinary incontinence in baseline and after 12 weeks of intervention;
  3. To evaluate the pelvic floor muscle functionality: To evaluate the pelvic floor muscle functionality, using PERFECT Scale and Pressure Biofeedback in baseline and after 12 weeks of intervention;
  Other Names: Pelvic Floor Muscle Training in group
  Arms: Experimental
Other: Control — 1. Profile of participants: an anamnesis file was used to collect personal data;
  2. To evaluate the quality of life: To evaluate the quality of life, using International Consultation on Incontinence Questionnaire (ICIQ-Short form) in women with urinary incontinence in baseline and after 12 weeks of intervention;
  3. To evaluate the pelvic floor muscle functionality: To evaluate the pelvic floor muscle functionality, using PERFECT Scale and Pressure Biofeedback in baseline and after 12 weeks of intervention;
  Other Names: Pelvic Floor at Home
  Arms: Control

SUMMARY:
Aim: To assess the influence of pelvic floor muscles group training in the quality of life and functionality of these muscles in women with UI.

Study design: This is a randomized controlled trial.

DETAILED DESCRIPTION:
Search location: Urogynecology Ambulatory Care of Porto Alegre Clinical Hospital (HCPA)

Patients or participants: Women will be included in aged 35-70 years who have had sexual intercourse in the last 12 months and who are able to understand the instruments, besides signing an informed consent form. Women will be excluded with latex allergy, who have made pelvic radiotherapy, or be undergoing chemotherapy, puerperal a year, or who use antidepressants and / or anxiolytics.

Intervention and measures: The evaluation consists of a medical history form, which will include personal data; the assessment of the MAP function is performed by the pressure biofeedback; for assessment of quality of life will use the questionnaire ICQI-SF and sexual function the PISQ-12 before and after Pelvic Floor Muscle Training.

Expected results: To estimate effectiveness of Pelvic Floor Muscle Training in the quality of life and functionality of these muscles in women with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Have urinary incontinence;
* Age between 35 and 70 years;
* Have sexual intercourse in the last 6 months;
* Participants should understand the instruments used in the research;
* Accept to participate in the study and sign the Term of Free and Informed Consent.

Exclusion Criteria:

* Latex allergy;
* Have performed or are undergoing pelvic radiotherapy;
* Be performing chemotherapy treatment;
* Women who delivered during the last 12 months;
* Have participated in individual or group MAP training in the last 6 months;
* Have contraction of the pelvic floor muscles grade zero (0).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Quality of life in women with urinary incontinence | 12 weeks
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) - scored between 0 and 21.

CONTACTS AND LOCATIONS:
Overall Officials: José Geraldo Lopes Ramos, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322